CLINICAL TRIAL: NCT01205412
Title: An Observational, Epidemiological Study on the Prevalence of Human Papillomavirus (HPV) Types in Women in the Kingdom of Bahrain
Brief Title: An Observational Study on the Prevalence of Human Papillomavirus Types in Women in the Kingdom of Bahrain
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112710
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endocervical samples

GROUPS / COHORTS (1):
- Assessed Cohort: Subjects attending out-patient health services for routine cervical screening or presenting for post-natal check up
  Interventions: Procedure: Endocervical samples

INTERVENTIONS:
Procedure: Endocervical samples — Endocervical samples collection during routine gynaecological examinations

SUMMARY:
The purpose of this study is to determine the Human Papillomavirus (HPV) prevalence and HPV type distribution among women ≥ 20 years of age attending routine cervical screening and among women ≥ 16 years of age presenting for post-natal check up in the Kingdom of Bahrain.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 20 years of age attending a clinic for routine cervical screening OR
* Women ≥ 16 years of age presenting for post-natal check-ups
* Women providing a cervical sample
* Written informed consent or oral-witnessed thumb printed informed consent obtained from the subject

Exclusion Criteria:

* Referral for abnormal cervical sample at the current visit
* Abundant menstrual bleeding or vaginal discharge not allowing appropriate screening to be performed (Note: Enrolment can be delayed until this condition is resolved)
* Pregnant women
* History of hysterectomy
* Known diagnosis of immunosuppression, or patient on immunosuppressives
* Having received one or more doses of human papillomavirus vaccine prior to participating in the study

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women ≥ 20 years of age, attending out-patient health services for routine cervical screening and women ≥ 16 years of age presenting for post-natal check up in the Kingdom of Bahrain.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of any Human Papillomavirus (HPV) deoxyribonucleic acid (DNA) and HPV type distribution among women undergoing cervical sample testing and post-natal check up. | Average time frame: 12 months

SECONDARY OUTCOMES:
Prevalence of any HPV DNA and HPV type distribution among women of different age strata undergoing cervical sample testing and post-natal check up. | Average time frame: 12 months
Behavioural risk factors | During visit 1 (day 0)
Awareness of HPV in relation to transmission and cause of cervical cancer | Average time frame: 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manama, Bahrain

REFERENCES:
- [Derived] Moosa K, Alsayyad AS, Quint W, Gopala K, DeAntonio R. An epidemiological study assessing the prevalence of human papillomavirus types in women in the Kingdom of Bahrain. BMC Cancer. 2014 Dec 3;14:905. doi: 10.1186/1471-2407-14-905. PMID 25466757